CLINICAL TRIAL: NCT01799005
Title: Impact of Dietary Flavanols on Vascular Health in a General Population of Healthy Middle-aged Europeans: a Randomized Controlled Study
Brief Title: FLAVIOLA Health Study
Acronym: FHS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Principal Investigator, Klinik für Kardiologie, Pneumologie und Angiologie, PD Dr. med. Christian Heiss, Heinrich-Heine University, Duesseldorf
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FHS
Record Dates: First submitted 2013-02-24; First posted 2013-02-26 (Estimated); Last update posted 2015-02-03 (Estimated); Status verified 2015-02

CONDITIONS: Vascular Health
Keywords: flavanols; diet; endothelial function; blood pressure; FLAVIOLA

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- flavanol rich intervention (Active Comparator): Ingestion of 410mg flavanols twice a day for 30 days
  Interventions: Dietary Supplement: Flavanol (410 mg)
- flavanol free intervention (Placebo Comparator): Ingestion of a macro and micro nutrients matched flavanol free drink
  Interventions: Dietary Supplement: Control (no flavanols)

INTERVENTIONS:
Dietary Supplement: Flavanol (410 mg)
  Other Names: Ingestion of intervention drink containing 410 mg flavanols twice a day for 30 days
  Arms: flavanol rich intervention
Dietary Supplement: Control (no flavanols)
  Other Names: Ingestion of a macro- and micronutrient matched control drink that is free of flavanols twice per day
  Arms: flavanol free intervention

SUMMARY:
Atherosclerosis progressively occurs with increasing age in the general population. So far most dietary intervention studies with flavanols were performed over short time frames and in small groups of young healthy and older patients with manifest cardiovascular disease, respectively. Vascular health is defined as absence of vascular disease and the presence of optimal parameters that determine the development and progression of arteriosclerosis (endothelial function, blood pressure, plasma lipids, and glucose). It is not clear whether flavanols can improve parameters of vascular health, most importantly endothelial function, when given repetitively to healthy middle aged and which factors affect the efficacy of flavanol interventions.

ELIGIBILITY:
Inclusion Criteria:

* male, age 35-60 years, healthy
* female, age 35-60 years, healthy

Exclusion Criteria:

* diabetes mellitus, acute inflammation, arrhythmia, active malignancy, terminal renal failure, signs, symptoms or medication indicative of manifest cardiovascular disease (CAD, PAD, CVD)

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-02; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Endothelial function | Time points: day 0 [baseline], and day 30 each 0 and 2h.

SECONDARY OUTCOMES:
Blood pressure | Time points: day 0 [baseline], and day 30 each 0 and 2h.
Glucose | Time points: day 0 [baseline], and day 30 each 0 and 2h.
Plasma lipids | Time points: day 0 [baseline], and day 30 each 0 and 2h.

OTHER OUTCOMES:
Flavanol metabolites | day 0 [baseline], and day 30 each 0 and 2h
Microparticles | Time points: day 0 [baseline], and day 30 each 0 and 2h.
Dietary pattern | Time points: day 0 [baseline] and day 30
Vascular stiffness | Time points: day 0 [baseline], and day 30 each 0 and 2h.
Microvascular function | Time points: day 0 [baseline], and day 30 each 0 and 2h.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Heiss, MD, Principal Investigator — Division of Cardiology, Pulmonology and Vascular Medicine; Malte Kelm, MD, Study Chair — Division of Cardiology, Pulmonology and Vascular Medicine
Locations (1):
- Division of Cardiology, Pulmonology and Vascular Medicine, Düsseldorf, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Sansone R, Rodriguez-Mateos A, Heuel J, Falk D, Schuler D, Wagstaff R, Kuhnle GG, Spencer JP, Schroeter H, Merx MW, Kelm M, Heiss C; Flaviola Consortium, European Union 7th Framework Program. Cocoa flavanol intake improves endothelial function and Framingham Risk Score in healthy men and women: a randomised, controlled, double-masked trial: the Flaviola Health Study. Br J Nutr. 2015 Oct 28;114(8):1246-55. doi: 10.1017/S0007114515002822. Epub 2015 Sep 9. PMID 26348767